CLINICAL TRIAL: NCT02375373
Title: Effects of Adding Chickpeas to the American Diet on Fecal Microbiota Composition and Markers of Inflammation
Brief Title: Effects of Adding Chickpeas to the American Diet (Long Term Study)
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: American Pulse Association (Other)
Responsible Party: Sponsor
Other Study IDs: 201400716 Long Term
Record Dates: First submitted 2015-02-24; First posted 2015-03-02 (Estimated); Results first posted 2016-02-19 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-01

CONDITIONS: Inflammation
Keywords: Gut Microbiota
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fecal
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational Chickpea Diet: Observed long-term to study legume intake and GI health (Observational Chickpea Diet)
  Interventions: Other: Observational Chickpea Diet

INTERVENTIONS:
Other: Observational Chickpea Diet — Individuals encouraged to maintain increased legume intake and explore new recipes that allow them to maintain a diverse menu of legume based foods.
  Fecal samples collected monthly.
  Other Names: Go'Bonzo's

SUMMARY:
This prospective study will assess the effects of adding legumes, especially chick peas, to the diet of healthy adults on the commensal bacteria from feces of human subjects and resulting self-reported GI symptoms as well as markers of immune function.

DETAILED DESCRIPTION:
Long-term observational study:

Subjects enrolled will participate in an observational setting for three months. During this time period, individuals will be encouraged, to maintain increased legume intake and explore new recipes that allow them to maintain a diverse menu of legume based foods. Fecal samples for microbiota analysis will be collected every month. Participants will record a weekly online questionnaire about legume intake and GI health as well as other health status updates. While participants will be encouraged to maintain regular intake of chickpeas throughout the long-term study, consumption of other legumes will be encouraged.

ELIGIBILITY:
Inclusion Criteria:

* Good Health
* No systemic antibiotics during the preceding two months
* No medication suppressing immune function
* Willingness to provide basic demographic as well as medical history data

Exclusion Criteria:

* Gastric Ulcers
* Inflammatory Bowel Disease (IBD) or Irritable Bowel Syndrome (IBS)
* Chronic constipation/diarrhea
* Body Mass Index (BMI) > 30
* Dietary restrictions that prevent legume intake
* Currently on any medication that can affect GI transit time
* Consumption of >3 servings/week of chickpeas or >6 servings/week of legumes BEFORE study begins

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals directly associated with the University of Florida (faculty, staff, students) or through the University of Florida's Health Street program.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2015-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Volker Mai, PhD, MPH, Principal Investigator — Associate Professor
Locations (1):
- Emerging Pathogens Institiute, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Obersvational Chickpea Diet: Observed long-term to study legume intake and GI health (Observational Chickpea Diet)
  Observational Chickpea Diet: Individuals encouraged to maintain increased legume intake and explore new recipes that allow them to maintain a diverse menu of legume based foods.
  Fecal samples collected monthly.
Period: Overall Study
Arm/Group | Obersvational Chickpea Diet
Started | 12
Completed | 1
Not Completed | 11
Not completed — Withdrawal by Subject | 11

BASELINE CHARACTERISTICS:
Arm/Group | Obersvational Chickpea Diet
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Changes in Number of 16S RNA Sequences on Days 31, Day 62, and Day 93.
Description: Compare the gut microbiota composition of individual subjects before and after the implementation of a controlled and observed diet of chickpeas and legume products.
Time Frame: Change from Day 31, Day 62, and Day 93
Population: Due to the rate of withdrawal from this study only one participant completed and this data was used for the outcome measures.
Measure: Mean (97.5% Confidence Interval); unit: sequences
Arm/Group | Obersvational Chickpea Diet
Number analyzed (Participants) | 1
sequences
  Day 31 | 49171 [49171 to 49171]
  Day 62 | 48925 [48925 to 48925]
  Day 93 | 49053 [49053 to 49053]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Obersvational Chickpea Diet
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No